CLINICAL TRIAL: NCT03050515
Title: Fecal Microbiota Transplantation for the Treatment of Recurrent Urinary Tract
Brief Title: Fecal Microbiota Transplantation for the Treatment of Recurrent Urinary Tract Infections
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Felicia Lane, Division Director of Female Pelvic Medicine and Reconstructive Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-3541
Record Dates: First submitted 2017-02-03; First posted 2017-02-13 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Recurrent Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fecal Transplant (Experimental): Enrolled and screened patients will receive a donor directed fecal transplant via retention enema. This procedure will take place at the University of California Irvine Women's Health Center on the day of the participant's choosing.
  The day prior to the procedure, the participant will undergo a bowel prep and stop all prophylactic antibiotics. On the day of procedure, the patient will present to the clinic and undergo a simple, retention enema. This procedure takes about 30-40 minutes to complete and does not require any anesthesia or sedation.
  Interventions: Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — This is a single arm study. All participants will receive a single fecal transplant to determine effectiveness in treating refractory recurrent urinary tract infections.
  Other Names: FMT; Fecal Transplant

SUMMARY:
Recurrent urinary tract infections are quickly becoming a public health obstacle in our aging population. Almost 50% of women have at least one urinary tract infection in their lifetime; following this first infection, there is a 25-35% chance that she will have another infection in the subsequent 3-6 months. With each documented infection, a patient receives anywhere from a three to seven day course of antibiotics for treatment. Repeated courses of antibiotics often lead to the development of multi-drug resistant infections that are difficult to treat with our arsenal of oral medications. It is theorized that most, if not all, urinary tract infections are caused by bacteria from the gastrointestinal tract. If there is a generalized gut dysbiosis due to repeated courses of oral antibiotics, it will likely be difficult to ever adequately treat repeat urinary tract infections. This same theory led to the development and utilization of fecal microbiota transplantation in the treatment of refractory Clostridium difficile diarrhea. There are now several studies that have reported on the efficacy of fecal transplantation in the treatment of C.difficile infections as well as the correction of gut dysbiosis. Given this positive response in treatment of refractory infectious diarrhea, the investigators propose that the correction of gut dysbiosis can also treat refractory recurrent urinary tract infections. Therefore, the investigators propose this pilot study to determine the effectiveness of fecal transplantation in the treatment of refractory, recurrent urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Meet criteria for recurrent urinary tract infections A. Each infection with bacterial colony count of greater than 100,000 AND B. 2 culture proven urinary tract infections within the preceding 6 months or culture proven urinary tract infections within the preceding 12 months
* Failed conservative management of recurrent urinary tract infections A. Completed 6-month trial of Macrobid, Trimethoprim or Methenamine suppression OR B. Completed 6-week series of intravesical instillations with DMSO or heparin/lidocaine

Exclusion Criteria:

* Pregnant
* Managed with a colostomy
* Managed with a suprapubic catheter
* Known renal abscess
* Acute or chronic renal failure
* Cardiac disease
* Rectal prolapse or bleeding
* Colon surgery in preceding 12 months

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-02-23 (Actual)

PRIMARY OUTCOMES:
Change in frequency of culture proven urinary tract infections following fecal transplant | 6 months
  Recurrent urinary tract infections are defined as 2 or more urine culture proven urinary tract infections in 6 months or 3 or more culture proven urinary tract infections in 12 months. To assess complete treatment success following fecal transplant, the investigators will collect urine cultures 1 month, 3 months and 6 months after fecal transplantation, as well as with any symptoms of a urinary tract infection, to determine the frequency of culture proven urinary tract infections over a 6 month time period following fecal transplant.

SECONDARY OUTCOMES:
Efficacy of fecal transplant in transforming recurrent urinary tract infection bacteria profile to that of pan-sensitive organisms on urine culture specimens | 6 months
  Often, patients with refractory recurrent urinary tract infection become infected with bacteria that are multi-drug resistant and therefore difficult to treat. To assess if a fecal transplant can alter the bacterial antibiotic susceptibility profile, the investigators will evaluate urine cultures 1 month, 3 months and 6 months after fecal transplant to test for infection and then to assess the antibiotic resistance profile.
Change in the gut microbiome following fecal transplantation measured via 16s sequencing of stool samples | 6 months
  The gut microbiome is an evolving field of research, especially following a fecal transplant. The investigators will collect a stool sample prior to fecal transplant and then at regular intervals following fecal transplant (1 day, 1 week, 1 month, 3 months and 6 months post-transplantation) to determine how a patient's gut microbiomes (via 16s sequencing) is affected by fecal transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Lane, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UCI Women's Healthcare Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeney SES, Avelar-Barragan J, Whiteson K, Chang J, Dutta S, Lane F. Fecal Putative Uropathogen Abundance and Antibiotic Resistance Gene Carriage in Women With Refractory Recurrent Urinary Tract Infection Treated With Fecal Microbiota Transplantation. Female Pelvic Med Reconstr Surg. 2022 Apr 1;28(4):213-219. doi: 10.1097/SPV.0000000000001090. Epub 2021 Oct 1. PMID 34608030